CLINICAL TRIAL: NCT04849702
Title: Comparison of the Clavien-Dindo and Comprehensive Complication Index Systems for Grading of Surgical Complications After Colorectal Resections.
Brief Title: Comparison of the Clavien-Dindo and Comprehensive Complication Index
Status: Completed | Type: Observational
Sponsor: Jessa Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2020007
Record Dates: First submitted 2021-04-02; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Complication of Surgical Procedure; Colorectal Disorders; Clavien Dindo; Comprehensive Complication Index

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Postoperative complication after colorectal resection: Documentation of all postoperative complications after colorectal resections
  Interventions: Procedure: No intervention was compared

INTERVENTIONS:
Procedure: No intervention was compared — No intervention was compared

SUMMARY:
Our aim was to compare 2 postoperative complication scoring systems in predicting length of hospital stay and in-hospital costs after colorectal resections.

DETAILED DESCRIPTION:
Introduction: Postoperative complications are associated with prolonged hospital stay and rise in costs of treatment. The Comprehensive Complication Index (CCI) was developed as a scoring system that does not only take the most severe complication into account, but all complications after surgery. Our aim was to compare the Clavien-Dindo scoring system with the CCI in predicting length of hospital stay (LOHS) and in-hospital costs after colorectal resections.

ELIGIBILITY:
Inclusion Criteria:

* Only patients that underwent a colorectal resection were included

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Data of patients in which complications occurring after surgical procedures, performed between October 2012 and September 2013, were recorded.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2012-10-20 (Actual); Primary Completion 2013-09-20 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | 1 year
Total in-hospital costs | 1 year

SECONDARY OUTCOMES:
Length of ICU stay | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Karel MC Smeyers, MD, Principal Investigator — Jessa hospital, Hasselt
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No